CLINICAL TRIAL: NCT04419051
Title: Owlet Band Observational Study: Observe the Use of a New Pregnancy Tracker for Expecting Mothers
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Owlet Baby Care, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: OWLB
Record Dates: First submitted 2020-02-20; First posted 2020-06-05 (Actual); Last update posted 2020-10-01 (Actual); Status verified 2020-09

CONDITIONS: Pregnancy; Anxiety; Stress
Keywords: Owlet; Pregnancy; Digital Health; Wellness
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Owlet Band — The Owlet Band is a wearable fabric band pregnancy tracker made up of small sensors that are able to detect natural low-level electrical signals normally produced by the mother's heart and baby's (fetal) heart.

SUMMARY:
This is an observational research study of a new pregnancy tracker used to gather information about a pregnant woman's general wellness.

DETAILED DESCRIPTION:
The Owlet Band is a wellness product (similar to a fitbit), it is not designed to be a "medical device". The study involves women age 18 and older who are currently pregnant, at least 24 weeks' gestation or later, and who live in the USA. Up to 8,000 pregnant women are expected to participate in the study. This study will involve review of Owlet Band data and participant responses to questionnaires throughout the study. The purpose of this research is to observe if using the new Owlet Band and the associated iPhone app can help pregnant women in managing their habits, anxiety, stress, enhancing bonding and attachment to their infant, while still maintaining their standard medical care.

ELIGIBILITY:
Inclusion Criteria:

* Must be at least 24 weeks pregnant with a singleton pregnancy
* Must be at least 18 years of age
* Must currently live in the United States
* Must have a compatible smartphone (Apple iOS Version 13 or above)
* Able to read and understand English in order to provide Informed Consent and follow study instructions

Exclusion Criteria:

* NA

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pregnant women 24 weeks' gestation and later
Sampling Method: Non-Probability Sample
Enrollment: 8000 (Estimated)
Dates: Start 2020-08-17 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Gather information | From date of enrollment until the date of reported delivery or early termination , whichever came first, assessed up to 16 weeks
  Successful collection of Owlet Band data from study participants
Gather information | Up to 16 weeks
  Completion of study questionnaires by at least 500 participants

SECONDARY OUTCOMES:
Management of anxiety State Trait Anxiety Inventory | Participant completion of the STAI questionnaire before wearing the Owlet Band and at Day 31 (+3 days)
  Change in anxiety as assessed by State Trait Anxiety Inventory (STAI)
Management of stress (Perceived Stress Scale) | Participant completion of the PSS questionnaire before wearing the Owlet Band and at Day 31 and Day 52 (+3 days)
  Change in perceived stress as assessed by Perceived Stress Scale (PSS)
Participant's experience while using the Owlet Band | Through study completion, up to 16 weeks
  Self-report of bonding and connection
Maintenance of standard medical care | Through study completion, up to 16 weeks
  Self-Report of standard medical care and unexpected or unscheduled visits

CONTACTS AND LOCATIONS:
Locations (1):
- Owlet Baby Care, Inc., Lehi, Utah, United States

IPD SHARING:
Plan to Share IPD: No